CLINICAL TRIAL: NCT02397785
Title: Treatment of Pain Using a Non-implanted Intra-vaginal Electrical Stimulation Device Compared to Sham Device in Chronic Pelvic Pain
Brief Title: Intra-vaginal Electrical Stimulation Device Compared to Sham Device for Chronic Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-150
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Pelvic Pain
Keywords: chronic pelvic pain; electrical stimulation; pelvic floor rehabilitation; neuromodulation
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ApexM Device (Experimental): InControl Medical created a line of products FDA approved for urinary incontinence and fecal incontinence (10). These devices are non-implanted, customizable, battery-operated vaginal probes made of medical grade silicon and provide electrical stimulation to the pelvic floor. One of the devices, ApexM™ provides electrical stimulation at frequencies alternating between 13 Hz and 50 Hz and allows the clinician to adjust the intensity as well as the duration of the electrical stimulation. The investigators propose the use of low power electrical stimulation for the treatment of pain in patients diagnosed with CPP. The electrical stimulation is delivered using ApexM™, adjusting the power to a sensory threshold to prevent muscle contraction.
  Interventions: Device: ApexM
- Sham Device (Sham Comparator): Subjects in the control arm will use a sham ApexM device. The original ApexM device will be modified to disable its electrical stimulation functionality. Otherwise, the devices are indistinguishable and possess identical dimensions. Although the sham device can be powered "on," the circuitry will be disconnected so that electrical stimulation is disabled.
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: ApexM — Subjects will apply conductive gel, insert the device to a minimum depth of 4 inches, and inflate until comfortably snug. The intensity is set exclusively by the physician to a tolerated sensory level, avoiding muscle contraction. At the target amplitude, patients will feel a non-painful fluttering or tapping sensation, Subjects will perform this for 6 sessions per week at 12 minutes per session for an additional 12 weeks. At each follow-up visit, investigators will re-evaluate the stimulation level and adjust to avoid muscle contraction.
  Other Names: pelvic electrical stimulation device
  Arms: ApexM Device
Device: Sham Device — Identical to ApexM but will not deliver any electrical stimulation
  Arms: Sham Device

SUMMARY:
The goal of the study is to evaluate the use of a personal intravaginal, non- implanted electrical stimulation device in the treatment of chronic pelvic pain. The investigators propose a randomized controlled trial comparing the investigated device to a sham device. The primary outcome is pain control using the visual analog scale and brief pain inventory (18). Hypothesis: Subjects will report increased pain relief with the electrical stimulation device compared to those using the sham device alone.

DETAILED DESCRIPTION:
Chronic pelvic pain (CPP) is a complex and devastating diagnosis, encompassing multiple different conditions. Many organ systems may be involved including musculoskeletal, neurologic, genitourinary, psychiatric or gastrointestinal systems. Furthermore, it can be associated with major insomnia, psychosexual trauma, and mood disorders resulting in challenging cases characterized by pain that is refractory to standard treatment modalities. In a study conducted by Mathias et al., one in seven women experience chronic pelvic pain. The economic burden can be substantial, with previous estimates of 2.8 billion dollars per year. (1) Dyspareunia is defined as recurrent or persistent pain associated with sexual intercourse and affects approximately 8-21% of women in the United States (19, 20). Understandably, women with dyspareunia often suffer a decline in sexual functioning. It may lead to decreased arousal, loss of libido, and anorgasmia. However, its impact extends beyond sexual functioning as it can affect a woman's reproductive health and overall sense of well-being. Previous estimates indicate that 88% of sexually active chronic pelvic pain patients report pain during or after intercourse (1).

Treatment of chronic pelvic is challenging due to a poor understanding of pain processing and physiology. Each patient's experience of pain is unique and may be any combination of visceral, neuropathic, or even somatic in etiology. Persistent pain despite aggressive treatment of organic etiologies may imply a psychogenic overlay. A comprehensive and integrative approach is ideal and may include physical therapy, medications, or cognitive behavioral therapy.

Pelvic floor physical therapy is an effective treatment. Pelvic floor rehabilitation addresses the pelvic floor dysfunction and may include manual therapy, transvaginal biofeedback and electrical stimulation. Reissing et al. performed a retrospective chart review and discovered that physical therapy, particularly internal manual techniques, is a successful technique in treating patients with vaginismus (5). Electrical stimulation (ES) to the pelvic floor is an effective treatment in vaginismus, vulvar vestibulitis, urinary urgency, and levator ani hypertonus (11-15). ES delivered specifically through a transcutaneous electrical nerve stimulator (TENS) unit results in notable benefit in pain and dyspareunia (8,12,21-23). Murina et al. conducted a randomized controlled trial comparing use of a vaginal probe delivering electrical stimulation to a sham device. In this study, they used a TENS unit to treat vestibulodynia using a protocol of 15 min of 10 Hz followed by 15 minutes of 50 Hz. These sessions were completed on a twice per week basis for 10 weeks. Pain scores, dyspareunia and overall sexual functioning were significantly improved in the active arm compared to placebo (8). Another study used a TENS unit to treat primary dysmenorrhea. In this protocol, the TENS unit was set to 100 Hz with 100ms pulse width for the first 8 hours of the menstrual cycle and then repeated for another menstrual cycle (9). A smaller study of 12 women used electrical stimulation biofeedback and gradual desensitization in the treatment of vaginismus. After treatment, all 12 women were able to have vaginal intercourse (13).

Electrical stimulation is used extensively for the treatment of various pain disorders. It is delivered through peripheral nerve stimulation, a TENS unit, or sacral neuromodulation using an implantable device. Electrical stimulation has three different programmable settings including the frequency, intensity and pulse duration. High frequency is considered as > 50 Hz whereas low frequency is < 10 Hz. The intensity, also known as the power, of the unit can be set to a sensory or motor threshold with any frequency (2).

There are several theories to explain the mechanism of action of electrical stimulation. TENS works by altering the ability to perceive pain signals. The gate theory is one proposed mechanism of action. Electrical stimulation of nerves via a specific dermatome results in a blocking or gating effect at the dorsal horn of the spinal cord. This inhibits the transmission of pain impulses to the upper nervous system. Also, low frequency stimulation of the dermatome can increase the level of endorphins, providing pain relief. (2) The sacral nerve roots 2-4 hold the autonomic and somatic innervation of the pelvic floor, bladder, and urethra. Therefore, stimulation of the sacral nerve roots 2-4 can provide a means to modulate impulses from the pelvic floor. Inhibition of afferent innervation from the pelvic floor or bladder is achieved with afferent activation of the sacral nerve roots using Interstim® or similar devices. In other words, stimulating the sacral nerve roots through neuromodulation has an inhibitory effect on pain pathways at the spinal cord level. (3) Treatment of chronic pelvic pain may include peripheral nerve stimulation via the posterior tibial nerve. This mixed nerve shares the same spinal origin as the innervation of the bladder and pelvic floor. Stimulation of the posterior tibial nerve travels retrograde to modulate the afferent input from the bladder or pelvic floor. (4) Therefore, it shares a similar mechanism of action to sacral neuromodulation but spares the patient the complications associated with surgical implantation of a device.

Despite its efficacy and benefits, electrical stimulation is time intensive and dependent upon a health care provider's schedule. It often causes the patient social embarrassment resulting in its inaccessibility. Although electrical stimulation provides pain relief, even highly motivated patients report that anxiety prohibits them from participation in physiotherapy (6). The investigators propose a novel treatment using a non-implanted intra-vaginal electrical stimulation device to be used in the comfort and privacy of the patient's home. This addresses several barriers associated with in office, standard pelvic floor physical therapy. Furthermore, a personal device allows the patient a more active role in her treatment, which can be empowering and ultimately, therapeutic.

InControl Medical created a line of products FDA approved for urinary incontinence and fecal incontinence (10). These devices are non-implanted, customizable, battery-operated vaginal probes made of medical grade silicon and provide electrical stimulation to the pelvic floor. One of the devices, ApexM™ provides electrical stimulation at frequencies alternating between 13 Hz and 50 Hz and allows the clinician to adjust the intensity as well as the duration of the electrical stimulation. The investigators propose the use of low power electrical stimulation for the treatment of pain in patients diagnosed with CPP. The electrical stimulation is delivered using ApexM™, adjusting the power to a sensory threshold to prevent muscle contraction.

The goal of the study is to evaluate the use of a personal intravaginal, non- implanted electrical stimulation device in the treatment of chronic pelvic pain. The investigators propose a randomized controlled trial comparing the investigated device to a sham device. The primary outcome is pain control using the visual analog scale and brief pain inventory (18). Hypothesis: Subjects will report increased pain relief with the electrical stimulation device compared to those using the sham device alone.

Secondary goals:

To evaluate the effect of ES on overall quality of life. Hypothesis: ES will improve quality of life as measured by the Short Form-36. (16) To evaluate the effect of ES on sexual function. Hypothesis: ES will improve sexual functioning as measured by Female Sexual Function Index (17) To evaluate the use of ES on use of pain medications. Hypothesis: ES will decrease dosage and frequency of pain medication use. This will be measured by use of a daily pain medication journal. Patients will complete a journal listing the type, amount and dosage of pain medications used on a daily basis.

SIGNIFICANCE If a positive effect is seen, a personal vaginal device designed for home use can be offered to patients with chronic pelvic pain. Patients would be able to take pelvic floor rehabilitation from the physical therapy office into their home. Furthermore, it would justify a larger, multi-center, randomized controlled trial comparing the ApexM™ device to standard in office physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Women >/= 18 years old who are sexually active or desire to be sexually active, no active infection, diagnosed with non-cyclic chronic pelvic pain, duration of symptoms greater than 6 months, neurologically intact, able to accommodate and tolerate the device, not pregnant and not attempting to achieve pregnancy.

Exclusion Criteria:

* Pregnancy, currently active in pelvic floor physical therapy, active malignancy, patients unable to contract their pelvic floor secondary to causes such as myelopathy, spinal cord trauma, patients with diabetes, vestibulodynia, vulvodynia, a pacemaker, defibrillator or other implanted neuro-modulatory devices, patients with a hypotonic pelvic floor, or those currently on treatment for pain with topical lidocaine, gabapentin or other medications or injections outside of standard analgesics, and severe psychiatric disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-04; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Uy-Kroh, MD, Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ApexM Device: InControl Medical created a line of products FDA approved for urinary incontinence and fecal incontinence. These devices are non-implanted, customizable, battery-operated vaginal probes made of medical grade silicone and provide electrical stimulation to the pelvic floor. The ApexM device provides electrical stimulation at frequencies alternating between 13 Hz and 50 Hz and allows the clinician to adjust the intensity as well as the duration of the electrical stimulation. Participants were instructed to apply conductive gel, insert the device to a minimum depth of 4 inches, and inflate until comfortably snug. The intensity was set exclusively by the physician to a tolerated sensory level, avoiding muscle contraction. Participants were instructed to complete 1 12-minute session at home per day, 6 days per week.
- Sham Device: Subjects in the control arm used a sham ApexM device. The original ApexM device was modified to disable its electrical stimulation functionality. Otherwise, the devices are indistinguishable and possess identical dimensions. Although the sham device can be powered "on," the circuitry was disconnected so that electrical stimulation is disabled. Participants were instructed to apply conductive gel, insert the device to a minimum depth of 4 inches, and inflate until comfortably snug. The intensity was set exclusively by the physician to a tolerated sensory level, avoiding muscle contraction. Participants were instructed to complete 1 12-minute session at home per day, 6 days per week.
Period: Overall Study
Arm/Group | ApexM Device | Sham Device
Started | 24 | 34
Completed | 22 | 25
Not Completed | 2 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ApexM Device | Sham Device | Total
Number analyzed (Participants) | 24 | 34 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (9.5) | 33.8 (10.5) | 33.2 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 34 | 58
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 20 | 30 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 34 | 58
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.0 (5.8) | 28.1 (6.3) | 27.6 (6.0)
Employment Status [Count of Participants; unit: Participants]
  Employed | 19 | 27 | 46
  Unemployed | 5 | 7 | 12
Annual Household Income [Count of Participants; unit: Participants]
  <$25,000 | 8 | 5 | 13
  $25,001-$50,000 | 4 | 8 | 12
  $50,001-$75,000 | 8 | 7 | 15
  $75,001-$100,000 | 1 | 5 | 6
  >$100,000 | 3 | 9 | 12
Highest Education Level Completed [Count of Participants; unit: Participants]
  < High School | 1 | 0 | 1
  High School / GED | 6 | 9 | 15
  College | 11 | 18 | 29
  Graduate/Professional Degree | 6 | 7 | 13
Total Parity [Count of Participants; unit: Participants]
  0 | 17 | 18 | 35
  1 | 2 | 6 | 8
  >=2 | 5 | 10 | 15
Vaginal Parity [Mean (Standard Deviation); unit: Vaginal Births] | 1.8 (1.2) | 1.1 (1.3) | 1.3 (1.2)
Menopausal Status [Count of Participants; unit: Participants]
  Pre-Menopausal | 21 | 30 | 51
  Post-Menopausal | 3 | 4 | 7
Pain Duration [Mean (Standard Deviation); unit: years] | 4.9 (3.4) | 11.0 (12.6) | 8.5 (10.3)
Endometriosis [Count of Participants; unit: Participants]
  Yes | 8 | 18 | 26
  No | 16 | 16 | 32
History of Pelvic Floor Physical Therapy [Count of Participants; unit: Participants]
  Yes | 4 | 9 | 13
  No | 20 | 25 | 45
History of Depression [Count of Participants; unit: Participants]
  Yes | 9 | 21 | 30
  No | 15 | 13 | 28
History of Sexual Abuse [Count of Participants; unit: Participants]
  Yes | 5 | 9 | 14
  No | 19 | 25 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain on the Visual Analog Scale (VAS) at Week 12
Description: The Visual Analog Scale assesses self-reported pain scores. Patients were asked to record their average pain over the past 4 weeks by placing an "X" on a 10-cm line, with 0 representing no pain and 100 representing the worst pain imaginable. Pain scores were determined by research personnel by measuring the distance (in mm) from 0 to the X. Change = (Week 12 Score - Baseline Score).
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 VAS scores available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 22 | 25
units on a scale | -8.5 (30.9) | -7.4 (25.0)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; It was calculated that 52 participants (26 in each arm) was sufficient to detect a 30% reduction in the VAS score (⍺ = 0.05, β = 0.80) from baseline to 12 weeks using paired t-tests, assuming average pain of 80-90 on the VAS and 10% drop-out. Because stratified randomization was performed on the basis of levator ani muscle spasm, there was an imbalance between the size of the sham and active groups, and 58 subjects were ultimately recruited with approval from the Institutional Review Board; Test type: Superiority; p = 0.8979, t-test, 2 sided

2. Secondary Outcome: Change From Baseline in Quality of Life on Short Form 36 (SF-36) Physical Functioning Scale
Description: Short Form-36 is a validated, self-reported instrument used to evaluate overall quality of life. The SF-36 consists of 8 sub-scales: 1) physical functioning, 2) role limitations due to physical health, 3) role limitations due to emotional problems, 4) energy/fatigue, 5) emotional well-being, 6) social functioning, 7) pain, 8) general health. Change = (Week 12 Score - Baseline Score). Scores for each sub-scale range from 0-100. Higher scores indicate better function / fewer symptoms.
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 SF-36 scores available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 22 | 25
units on a scale | 1.4 (4.1) | 1.6 (13.9)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Superiority; p = 0.9338, Sign test

3. Secondary Outcome: Change From Baseline in Quality of Life on Short Form 36 (SF-36) Role Limitations Due to Physical Health Scale
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 SF-36 scores available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 22 | 25
units on a scale | 1.13 (50.9) | 21 (43.7)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Superiority; p = 0.1568, Sign test

4. Secondary Outcome: Change From Baseline in Quality of Life on Short Form 36 (SF-36) Role Limitations Due to Emotional Problems Scale
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 SF-36 scores available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 22 | 25
units on a scale | -7.6 (43.5) | 2.7 (35.9)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Superiority; p = 0.3817, Sign test

5. Secondary Outcome: Change From Baseline in Quality of Life on Short Form 36 (SF-36) Energy/Fatigue Scale
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 SF-36 scores available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 22 | 25
units on a scale | 1.8 (19.1) | 7.2 (15.0)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Superiority; p = 0.2860, Sign test

6. Secondary Outcome: Change From Baseline in Quality of Life on Short Form 36 (SF-36) Emotional Wellbeing Scale
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 SF-36 scores available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 22 | 25
units on a scale | -2.9 (12.3) | 0.8 (11.4)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Superiority; p = 0.2884, Sign test

7. Secondary Outcome: Change From Baseline in Quality of Life on Short Form 36 (SF-36) Social Function Scale
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 SF-36 scores available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 22 | 25
units on a scale | -3.4 (15.5) | 5.5 (18.8)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Superiority; p = 0.0855, Sign test

8. Secondary Outcome: Change From Baseline in Pain on Short Form 36 (SF-36) Pain Scale
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 SF-36 scores available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 22 | 25
units on a scale | 5.2 (21.9) | 18.1 (17.1)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Superiority; p = 0.0287, Sign test

9. Secondary Outcome: Change From Baseline in Quality of Life on Short Form 36 (SF-36) General Health Scale
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 SF-36 scores available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 22 | 25
units on a scale | -3.1 (9.9) | 0 (10)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Superiority; p = 0.2887, Sign test

10. Secondary Outcome: Change From Baseline in Pain on Brief Pain Inventory (BPI) Pain Severity Scale
Description: The Brief Pain Inventory (BPI) is a validated, self-reported instrument used to evaluate pain symptoms within the last 24 hours. The BPI consists of 2 sub-scales: 1) pain severity, 2) pain interference. Change = (Week 12 Score - Baseline Score). Scores for each sub-scale range from 0-10. Lower scores indicate better function / fewer symptoms.
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 BPI scores available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 22 | 25
units on a scale | -0.4 (2.3) | -0.4 (1.5)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Superiority; p = 0.9954, Sign test

11. Secondary Outcome: Change From Baseline in Pain on Brief Pain Inventory (BPI) Pain Interference Scale
Description: as for outcome 10
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 BPI scores available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 22 | 25
units on a scale | -0.06 (3.2) | -1.1 (2.0)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Superiority; p = 0.0574, Sign test

12. Secondary Outcome: Change From Baseline in Quality of Life on Female Sexual Function Index (FSFI) Scale
Description: The Female Sexual Function Index is a validated, self-reported instrument used to evaluate sexual function and symptoms. The FSFI consists of 6 sub-scales: 1) desire [score range = 1.2 - 6], 2) arousal [score range = 0 - 6], 3) lubrication [score range = 0 - 6], 4) orgasm [score range = 0 - 6], 5) satisfaction [score range = 0 - 6], 6) pain [score range = 0 - 6]. The full FSFI consists of 19 questions, and the total score ranges from 1.2 - 36. Change = (Week 12 Score - Baseline Score). Higher scores indicate better function / fewer symptoms.
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 FSFI scores available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 22 | 25
units on a scale | 2.7 (8.0) | 1.9 (9.2)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Superiority; p = 0.7827, Sign test

13. Secondary Outcome: Change From Baseline in Quality of Life on Pelvic Floor Distress Inventory (PFDI) Pelvic Organ Prolapse Distress Inventory (POPDI) Sub-Scale
Description: The Pelvic Floor Distress Inventory is a 20-question, validated, self-reported instrument used to evaluate pelvic floor symptoms. It consists of an overall scale (range: 0-300) comprised of 3 sub-scales: 1) Pelvic Organ Prolapse Distress Inventory (range: 0-100), 2) Colorectal Anal Distress Inventory (range: 0-100), and 3) Urinary Distress Inventory (range: 0-100). Change = (Week 12 Score - Baseline Score). Lower scores indicate better function / fewer symptoms.
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 PFDI scores available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 22 | 25
units on a scale | -4.7 (11.7) | -9.3 (13.0)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Superiority; p = 0.2114, Sign test

14. Secondary Outcome: Change From Baseline in Quality of Life on Pelvic Floor Distress Inventory (PFDI) Colorectal Anal Distress Inventory (CRADI) Sub-Scale
Description: as for outcome 13
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 PFDI scores available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 22 | 25
units on a scale | -4.1 (8.6) | -6.5 (14.2)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Superiority; p = 0.4986, Sign test

15. Secondary Outcome: Change From Baseline in Quality of Life on Pelvic Floor Distress Inventory (PFDI) Urinary Distress Inventory (UDI) Sub-Scale
Description: as for outcome 13
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 PFDI scores available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 22 | 25
units on a scale | -6.3 (17.6) | -10 (16.3)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Superiority; p = 0.4610, Sign test

16. Secondary Outcome: Change From Baseline in Quality of Life on Pelvic Floor Distress Inventory (PFDI) Total Scale
Description: as for outcome 13
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 PFDI scores available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 22 | 25
units on a scale | -15.2 (28.8) | -25.8 (33.9)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Superiority; p = 0.2556, Sign test

17. Secondary Outcome: Change From Baseline in Weekly Ibuprofen Use
Description: Patients were asked to record weekly doses of over-the-counter pain medications taken, including ibuprofen (mg), naprosyn (mg), acetaminophen (mg), and opioids (calculated morphine equivalents). Change = (Week 12 total - Week 1 total).
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 medication diaries available.
Measure: Mean (Standard Deviation); unit: mg/week
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 20 | 21
mg/week | 200 (836) | -400 (1201)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Superiority; p = 0.0723, t-test, 2 sided

18. Secondary Outcome: Change From Baseline in Weekly Naprosyn Use
Description: as for outcome 17
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 medication diaries available.
Measure: Mean (Standard Deviation); unit: mg/week
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 20 | 21
mg/week | -35.3 (250) | -62.9 (288)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Superiority; p = 0.7456, t-test, 2 sided

19. Secondary Outcome: Change From Baseline in Weekly Acetaminophen Use
Description: as for outcome 17
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 SF-36 scores available.
Measure: Mean (Standard Deviation); unit: mg/week
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 20 | 21
mg/week | 125 (559) | -333 (1238)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Superiority; p = 0.1380, t-test, 2 sided

20. Secondary Outcome: Change From Baseline in Weekly Opioid Use
Description: as for outcome 17
Time Frame: Baseline and Week 12
Population: Based on the intention-to-treat population. All participants with Baseline and Week 12 SF-36 scores available.
Measure: Mean (Standard Deviation); unit: morphine equivalents/week
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 20 | 21
morphine equivalents/week | -0.25 (1.1) | 0 (0)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Superiority; p = 0.3155, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the entire study period for each participant (12 weeks). Following study completion, participants were encouraged to contact the researchers in the event of any future device-related adverse outcome, and they were offered assistance in scheduling follow-up visits with the Chronic Pelvic Pain Center at our institution.
Description: Adverse event reporting was conducted through use of standardized questions asked at the time of each trial visit (every 4 weeks). Additionally, participants were given contact information for multiple methods of reporting adverse events, including contact information for the researchers, the general research nurse office, the on-call gynecologist, and the Institutional Review Board.
Arm/Group | ApexM Device | Sham Device
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/34
Other Adverse Events (participants affected / at risk) | 14/24 | 4/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ApexM Device (N=24) | Sham Device (N=34)
Vaginal Discharge (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Tingling Sensation (Product Issues) | 8 (8) | 0 (0) — Resolved with device repositioning and further instruction/teaching about correct positioning
Pelvic Cramping (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 2 (2) | 0 (0)
Vaginal Soreness (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT02397785/Prot_SAP_000.pdf